CLINICAL TRIAL: NCT03935217
Title: Multi-center, Prospective, Randomized, Placebo-Controlled, Delayed Treatment, Double-Blind Study to Evaluate the Effectiveness and Safety of a Single Oral Dose of Solosec® for the Treatment of Trichomoniasis
Brief Title: A Phase 3 Study of Solosec® for the Treatment of Trichomoniasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lupin Research Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SEC-WH-301
Record Dates: First submitted 2019-04-30; First posted 2019-05-02 (Actual); Results first posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Trichomonas Infection
Keywords: Vaginal Itching; Vaginal Discharge
MeSH Terms: conditions — Trichomonas Infections; Vaginal Discharge | interventions — secnidazole

STUDY DESIGN:
Intervention Model Description: For primary phase of study, patients were randomly assigned in a 1:1 ratio to either Solosec or Placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Solosec (containing 2 grams of secnidazole) (Experimental): Orally administered as a single dose with applesauce.
  Interventions: Drug: Secnidazole
- Placebo (Placebo Comparator): Orally administered as a single dose with applesauce.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Secnidazole — Oral Granules containing secnidazole
  Other Names: Solosec®
  Arms: Solosec (containing 2 grams of secnidazole)
Drug: Placebo — Oral Granules of placebo manufactured to mimic secnidazole
  Arms: Placebo

SUMMARY:
This is a Phase 3, multi-center, prospective, randomized, placebo-controlled, delayed treatment, double-blind, study to evaluate the effectiveness, and safety of a single, oral dose of Solosec® containing 2 grams of secnidazole in female patients with trichomoniasis.

DETAILED DESCRIPTION:
The study will consist of a primary study phase (Visit 1 (baseline) to Visit 2 (Day 6-12)) and a follow-up phase (Visit 2 to Visit 3 (7-12 days post Visit 2)). During the primary phase patients will be randomly assigned in a 1:1 ratio to either Solosec or placebo. Patients will return to the clinic for the "test of cure" (TOC) visit to be conducted on Days 6-12 (Visit 2).

To ensure all patients receive treatment and to maintain the double-blind, after completion of the primary phase, patients will receive the opposite treatment , (placebo patients will receive Solosec and vice versa). Patients with V2 cultures that are subsequently positive for T. vaginalis will return to the clinic for Visit 3 (V3) assessments and investigator assessment of need for additional therapy (an additional Visit 4 may be scheduled at the investigator's discretion if culture at V3 is positive).

Summary of results includes data reported during the primary phase of the study [Visit 1 (baseline) to Visit 2/TOC (Day 6-12)]

ELIGIBILITY:
Inclusion Criteria:

* adult female or post-menarche adolescent girl ≥12 years of age in general good health
* Have a diagnosis of trichomoniasis at the screening visit as determined by one of the following:

  * positive T. vaginalis NAAT test within 30 days of screening for which treatment has not been initiated.
  * positive OSOM® rapid test.
  * positive wet mount assessment.
* Agree to abstain from vaginal intercourse until the final study visit
* Agree not to have any vaginal penetration or use of any vaginal products for the duration of the study

Exclusion Criteria:

* Are pregnant, lactating, or planning to become pregnant during the study.
* Are suspected clinically (or confirmed diagnostically) of having alternative causes of vaginal symptoms including symptomatic vulvovaginal candidiasis, chlamydia, gonorrhea, or an active genital herpes outbreak
* Are suspected clinically of having an acute urinary tract infection.
* Have active genital lesions, including primary syphilitic chancres and herpes simplex virus lesions, or other vaginal or vulvar conditions which could confound the interpretation of the clinical response, as determined by the Investigator (patients with genital warts may be enrolled).
* Have received systemic antibacterial therapy or topical antimicrobial/antifungal/ immunomodulatory therapies in the genital area (vagina, vulva and surrounding soft tissue), within 14 days prior to the Baseline Visit (Day 1).

Min Age: 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Must be female
Enrollment: 147 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2020-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jackie Shaw, Study Director — Director, Clinical Operations
Locations (11):
- United States (11):
  - Site 1007, Birmingham, Alabama
  - Site 1003, North Miami, Florida
  - Site 1014, Chicago, Illinois
  - Site 1013, Jackson, Mississippi
  - Site 1009, Lawrenceville, New Jersey
  - Site 1008, Chapel Hill, North Carolina
  - Site 1004, Fayetteville, North Carolina
  - Site 1011, Charleston, South Carolina
  - Site 1001, Memphis, Tennessee
  - Site 1002, Memphis, Tennessee
  - Site 1006, Virginia Beach, Virginia

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: After publication of the primary study results, the research team will prepare final research data files that may be shared with other investigators, upon request.
Access Criteria: Requests for research data must be submitted to author CAM in writing, via a standard data request form, with a justification for how the data will be used. Author CAM and Lupin Pharmaceuticals will review all requests for research data obtained from this study. The mechanism by which the data will be made available to investigators will follow all NIH guidelines for data sharing as they evolve. At a minimum this would consist of a data use agreement that provides for commitments to use the data for research purposes only, secure the data with appropriate computer technology, obtain IRB approval, and destroy (or return) the data after analyses are complete.

REFERENCES:
- [Derived] Muzny CA, Van Gerwen OT, Kaufman G, Chavoustie S. Efficacy of single-dose oral secnidazole for the treatment of trichomoniasis in women co-infected with trichomoniasis and bacterial vaginosis: a post hoc subgroup analysis of phase 3 clinical trial data. BMJ Open. 2023 Aug 7;13(8):e072071. doi: 10.1136/bmjopen-2023-072071. PMID 37550019
- [Derived] Muzny CA, Schwebke JR, Nyirjesy P, Kaufman G, Mena LA, Lazenby GB, Van Gerwen OT, Graves KJ, Arbuckle J, Carter BA, McMahon CP, Eder S, Shaw J, Pandey B, Chavoustie SE. Efficacy and Safety of Single Oral Dosing of Secnidazole for Trichomoniasis in Women: Results of a Phase 3, Randomized, Double-Blind, Placebo-Controlled, Delayed-Treatment Study. Clin Infect Dis. 2021 Sep 15;73(6):e1282-e1289. doi: 10.1093/cid/ciab242. PMID 33768237

RESULTS

PARTICIPANT FLOW:
Groups:
- Solosec 2 Grams: Orally administered as a single dose with applesauce.
  Secnidazole: Oral Granules containing secnidazole
Period: Overall Study
Arm/Group | Solosec 2 Grams | Placebo
Started | 74 | 73
Completed | 73 | 70
Not Completed | 1 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Solosec 2 Grams: Orally administered as a single dose with applesauce.
  Secnidazole: Oral Granules containing secnidazole then
- Placebo: Orally administered as a single dose with applesauce.
  Placebo: Oral Granules of placebo manufactured to mimic secnidazole then
- Total: Total of all reporting groups
Arm/Group | Solosec 2 Grams | Placebo | Total
Number analyzed (Participants) | 74 | 73 | 147
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 74 | 72 | 146
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.5 (0) | 38.6 (0) | 37.6 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 73 | 147
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 72 | 71 | 143
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 68 | 66 | 134
  White | 4 | 6 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 74 | 73 | 147
Number of Participants for Modified intent to treat population [Count of Participants; unit: Participants] | 64 | 67 | 131

OUTCOME MEASURES:

1. Primary Outcome: Microbiological Cure at the TOC Visit
Description: Vaginal Culture negative for T. vaginalis at TOC Visit
Time Frame: Study Day 6-12
Population: Modified Intent to Treat Population (Patients with culture positive for T. vaginalis at baseline)
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Orally administered as a single dose with applesauce.
  Secnidazole: Oral Granules containing secnidazole
Arm/Group | Solosec 2 Grams | Placebo
Number analyzed (Participants) | 64 | 67
Participants | 59 | 1

ADVERSE EVENTS:
Time Frame: Data includes AEs reported during the primary phase of study [Visit 1 (baseline) to TOC/Visit 2 (day 6-12)] for each study patient.
Description: Adverse Event data reported for primary phase of study only. Subjects received either Solosec or Placebo (1:1) during primary phase of study.
Arm/Group | Solosec (Containing 2 Grams of Secnidazole) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/73
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/73
Other Adverse Events (participants affected / at risk) | 6/74 | 14/73
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Solosec (Containing 2 Grams of Secnidazole) (N=74) | Placebo (N=73)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Vulvovagnial candidiasis (Infections and infestations) | 2 (2) | 0 (0)
Trichomoniasis (Infections and infestations) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 5 (5)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-03-29): https://cdn.clinicaltrials.gov/large-docs/17/NCT03935217/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-20): https://cdn.clinicaltrials.gov/large-docs/17/NCT03935217/SAP_001.pdf